CLINICAL TRIAL: NCT04673344
Title: Collagen Scaffold Augmentation of High Grade Partial Rotator Cuff Tendon Tears Improves Early Functional Recovery: A Randomized Controlled Trial.
Brief Title: Regeneten Patch vs Standard Care in Partial Thickness Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTJO2020-0876
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Rotator Cuff Tears; Shoulder Surgery
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Partial Rotator Cuff Repair (No Intervention): Routine partial rotator cuff repair
- Partial Rotator Cuff Repair with Regeneten Scaffold (Active Comparator): Routine partial rotator cuff repair with the addition of the Regeneten scaffolding patch
  Interventions: Device: Regeneten Collagen Patch

INTERVENTIONS:
Device: Regeneten Collagen Patch — Partial rotator cuff repair surgery with the addition of the Regeneten scaffold
  Arms: Partial Rotator Cuff Repair with Regeneten Scaffold

SUMMARY:
Shoulder pain is a common complaint with the most common reason being tendinopathy and/or tearing of the rotator cuff. While many rotator cuff tears are often considered normal, age-related degenerative disorders, with either partial- or full-thickness rotator cuff tears evident in 4% of patients aged <40 years and in 54% of patients aged >60 years, once they become symptomatic and conservative management fails, they are typically repaired surgically. Data suggest that the incidence of surgery to repair and re-attach the cuff continues to rise. However, despite positive clinical results overall, reports of repair failure after surgery can range from 16%-94%, and of those that do fail, or fail to heal, generally do so within the first 3 to 6 months post-surgery.

Given the aforementioned reported issues with the gold standard for the treatment of unresponsive and symptomatic partial or full rotator cuff tears (surgical repair), together with the invasiveness of this surgery and lengthy period of restricted activity, other means of treatment have been proposed.

The REGENETEN scaffold/implant seeks to support new tendon growth and disrupt disease progression. This study seeks to investigate the outcome of surgical rotator cuff repair versus scaffold augmentation (using the REGENETEN scaffold) for symptomatic partial thickness rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 40-75 years with a partial-thickness rotator cuff tear (50% or more) confirmed on MRI scan that, in combination with patient-report symptoms and clinical examination by the orthopaedic surgeon, would confirm the rotator cuff tear as the primary pathology driving pain, symptoms and functional disability .
* Symptoms > 3 months
* Unsuccessful conservative treatment comprising of a corticosteroid injection (into the subacromial bursa) and physiotherapy (while it is acknowledged that a range of modalities may be available to patient's presenting with apparent symptomatic rotator cuff pathology, for the current study, physiotherapy has been defined specifically as a course of 'exercise-based' therapy specific to the individual patient, though generally comprising of exercises designed to strengthen the rotator cuff and scapula stabilizing musculature, improving flexibility and shoulder mobility)

Exclusion Criteria:

* Revision surgery
* Cervical pathology
* Adhesive capsulitis
* Multi-tendon tears
* Concomitant upper limb pathology (eg: arthritis, nerve compression)
* Infection
* Previous fracture
* Instability
* Pregnancy and lactation
* Professional athlete
* Worker's compensation or compensable claim
* Substance abuse or current mental illness
* Smoker
* Adverse reaction to bovine derived products

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rotator Cuff Healing | 24 months
  The status of rotator cuff healing as demonstrated on post-operative MRI (at 6, 12 and 24 months)
Participant Satisfaction: ASES assessment | 24 months
  Participant Satisfaction with their surgical outcomes will be measured with the use of the American Shoulder and Elbow Surgeons at 6 week, 3-, 6-, 12- and 24 months after surgery
Participant Satisfaction: WORC assessment | 24 months
  Participant Satisfaction with their surgical outcomes will be measured with the use of the Western Ontario Rotator Cuff Index at 6 week, 3-, 6-, 12- and 24 months after surgery
Participant Satisfaction: SANE assessment | 24 months
  Participant Satisfaction with their surgical outcomes will be measured with the use of the Single Assessment Numeric Evaluation at 6 week, 3-, 6-, 12- and 24 months after surgery
Participant Satisfaction: VR-12 assessment | 24 months
  Participant Satisfaction with their surgical outcomes will be measured with the use of the Veteran's Rand 12 assessment at 6 week, 3-, 6-, 12- and 24 months after surgery
Participant Satisfaction: GRC assessment | 24 months
  Participant Satisfaction with their surgical outcomes will be measured with the use of the Global Rating of Change scale at 6 week, 3-, 6-, 12- and 24 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States